CLINICAL TRIAL: NCT06919692
Title: Impact of Maternal Left-Lateral Recumbent Positioning in Pregnancies With Fetal Growth Restriction
Brief Title: Maternal Left Lateral Position in Fetal Growth Restriction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-0289
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Fetal Growth Restriction
Keywords: fetal growth restriction; left lateral position; maternal fetal medicine
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The sonographer doing the fetal biometry at enrollment and during the 4-week follow-up visit will be masked to the study group assigned to the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group A (Experimental): Pregnant persons randomized into this group will be instructed to practice left-lateral recumbent position for a period of 4-hours (cumulatively) daily for 4-weeks after enrollment. The participants will be advised to stretch for 10 mins after every hour of recumbent position. A per-protocol recommendation of mild to moderate intensity exercise 2-3 times a week will be advised. A healthy diet will also be recommended. The activity at home will be recorded via a smart watch.
  Interventions: Behavioral: Left lateral recumbent positioning
- Intervention group B (No Intervention): Pregnant persons in this group will continue to receive the 'standard of care', per clinical protocol. A recommendation of mild to moderate intensity exercise 2-3 times a week will be advised. A healthy diet will be recommended. The activity status at home will be recorded via a smart watch.

INTERVENTIONS:
Behavioral: Left lateral recumbent positioning — Left-lateral position is the recommended position of resting in pregnancy. The participants in the intervention group will be advised to practice this position with an intermittent 10-minute stretching after every hour of resting, with no more than 4-hours of this intervention per day.
  Arms: Intervention group A

SUMMARY:
The goal of this clinical trial is to learn if maternal left-lateral positioning in pregnancy works to treat fetal growth restriction. This study will also help us learn about the effects of left-lateral positioning on maternal metabolomics, maternal mental health, fetal cardiac function, and delivery outcomes. The main questions it aims to answer are:

* Does maternal left-lateral position in a pregnancy with fetal growth restriction improve the baby's growth?
* How are maternal metabolomics, delivery outcomes, maternal mental health, and fetal cardiac function impacted by maternal left-lateral position? Researchers will compare the intervention group to pregnancies with fetal growth restriction that receive standard of care (without left-lateral positioning) to see if left-lateral position improves fetal biometry in fetal growth restriction.

Participants will:

* Practice left-lateral position every day for 4 hours (cumulatively) with 10-mins stretching after every hour of left-lateral position, or continue to receive standard of care
* Visit the clinic once after 4 weeks for a follow-up research visit, and at the time of delivery

Tracking of the physical activity and adherence to left-lateral position at home in intervention group A will be done through a fitbit (smart watch) given during enrollment. A fitbit will also be given to participants in intervention group B, receiving standard of care, to monitor their physical activity trends at home.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant persons between 18 - 65 years of age, with a diagnosis of fetal growth restriction, with an estimated fetal weight less than tenth percentile
* Participants with a singleton pregnancy between 24- and 34-weeks' gestational age
* Participants with fluency in English or Spanish language

Exclusion Criteria:

* Patients with a known history of deep vein thrombosis, pulmonary embolism, or hypercoagulability disorder
* Patients with a pre-pregnancy BMI greater than 40
* Pregnancy with severe abnormality in umbilical artery Doppler flow, including absent end-diastolic flow (AEDF) and reverse end-diastolic flow (REDF)
* Patients receiving anticoagulation therapy
* Pregnancy with suspected chromosomal anomalies or a multifetal pregnancy
* Patients with an active smoking status during pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
Fetal biometry | 4 weeks after enrollment
  Fetal estimated fetal weight and abdominal circumference will be assessed and compared to enrollment values

SECONDARY OUTCOMES:
Fetal cardiac function | 4 weeks after enrollment
  Variables of fetal cardiac function including cardiac contractility and cardiac size and shape will be assessed using speckle tracking
Feto-Maternal Doppler flow | 4 weeks after enrollment
  Measures of Doppler flow including umbilical artery, middle cerebral artery, umbilical vein flow, and cerebroplacental ratio will be assessed
Delivery outcomes | At delivery
  Variables including gestational age at delivery, birthweight, neonatal arterial pH, APGAR scores, mode of delivery, indication of cesarean delivery, if applicable, will be recorded
Maternal Mental Health evaluation | 4 weeks after enrollment, and after delivery
  Maternal mental health assessment will be done via Edinburg Postnatal Depression Scale questionnaire. Based on questionnaire responses, participant will receive a score within range 0-30. A score of 10 or higher would require further evaluation for depression.
Maternal Metabolomics assessment | 4 weeks after enrollment, and after delivery
  Maternal metabolomics will be evaluated and compared to baseline via a blood and a urine sample at the 4-week follow-up and via a cord blood and a maternal blood sample at the time of delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Manesha Putra, MD, Principal Investigator — University of Colorado Anschutz, Department of Obstetrics and Gynecology
Locations (2):
- United States (2):
  - UCHealth Prenatal Diagnosis and Genetics Clinic - Anschutz Medical Campus, Aurora, Colorado
  - CU John C. Hobbins Perinatal Center, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics and the Society forMaternal-FetalMedicin. ACOG Practice Bulletin No. 204: Fetal Growth Restriction. Obstet Gynecol. 2019 Feb;133(2):e97-e109. doi: 10.1097/AOG.0000000000003070. PMID 30681542
- [Background] Gardosi J, Madurasinghe V, Williams M, Malik A, Francis A. Maternal and fetal risk factors for stillbirth: population based study. BMJ. 2013 Jan 24;346:f108. doi: 10.1136/bmj.f108. PMID 23349424
- [Background] Lees CC, Romero R, Stampalija T, Dall'Asta A, DeVore GA, Prefumo F, Frusca T, Visser GHA, Hobbins JC, Baschat AA, Bilardo CM, Galan HL, Campbell S, Maulik D, Figueras F, Lee W, Unterscheider J, Valensise H, Da Silva Costa F, Salomon LJ, Poon LC, Ferrazzi E, Mari G, Rizzo G, Kingdom JC, Kiserud T, Hecher K. Clinical Opinion: The diagnosis and management of suspected fetal growth restriction: an evidence-based approach. Am J Obstet Gynecol. 2022 Mar;226(3):366-378. doi: 10.1016/j.ajog.2021.11.1357. Epub 2022 Jan 10. PMID 35026129
- [Background] Baschat AA, Galan HL, Lee W, DeVore GR, Mari G, Hobbins J, Vintzileos A, Platt LD, Manning FA. The role of the fetal biophysical profile in the management of fetal growth restriction. Am J Obstet Gynecol. 2022 Apr;226(4):475-486. doi: 10.1016/j.ajog.2022.01.020. PMID 35369904
- [Background] DeVore GR, Gumina DL, Hobbins JC. Assessment of ventricular contractility in fetuses with an estimated fetal weight less than the tenth centile. Am J Obstet Gynecol. 2019 Nov;221(5):498.e1-498.e22. doi: 10.1016/j.ajog.2019.05.042. Epub 2019 May 30. PMID 31153929
- [Background] DeVore GR, Polanco B, Lee W, Fowlkes JB, Peek EE, Putra M, Hobbins JC. Maternal rest improves growth in small-for-gestational-age fetuses (<10th percentile). Am J Obstet Gynecol. 2025 Jan;232(1):118.e1-118.e12. doi: 10.1016/j.ajog.2024.04.024. Epub 2024 May 21. PMID 38842845
- [Background] Higuchi H, Takagi S, Zhang K, Furui I, Ozaki M. Effect of lateral tilt angle on the volume of the abdominal aorta and inferior vena cava in pregnant and nonpregnant women determined by magnetic resonance imaging. Anesthesiology. 2015 Feb;122(2):286-93. doi: 10.1097/ALN.0000000000000553. PMID 25603203
- [Background] Lee SW, Khaw KS, Ngan Kee WD, Leung TY, Critchley LA. Haemodynamic effects from aortocaval compression at different angles of lateral tilt in non-labouring term pregnant women. Br J Anaesth. 2012 Dec;109(6):950-6. doi: 10.1093/bja/aes349. Epub 2012 Oct 11. PMID 23059960
- [Background] Nelson DB, Stewart RD, Matulevicius SA, Morgan JL, McIntire DD, Drazner M, Cunningham FG. The Effects of Maternal Position and Habitus on Maternal Cardiovascular Parameters as Measured by Cardiac Magnetic Resonance. Am J Perinatol. 2015 Dec;32(14):1318-23. doi: 10.1055/s-0035-1563719. Epub 2015 Sep 16. PMID 26375044
- [Background] Laurin J, Persson PH. The effect of bedrest in hospital on fetal outcome in pregnancies complicated by intra-uterine growth retardation. Acta Obstet Gynecol Scand. 1987;66(5):407-11. doi: 10.3109/00016348709022043. PMID 3321864
- [Background] Palacio M, Mottola MF. Activity Restriction and Hospitalization in Pregnancy: Can Bed-Rest Exercise Prevent Deconditioning? A Narrative Review. Int J Environ Res Public Health. 2023 Jan 13;20(2):1454. doi: 10.3390/ijerph20021454. PMID 36674214
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; Lauder J, Sciscione A, Biggio J, Osmundson S. Society for Maternal-Fetal Medicine Consult Series #50: The role of activity restriction in obstetric management: (Replaces Consult Number 33, August 2014). Am J Obstet Gynecol. 2020 Aug;223(2):B2-B10. doi: 10.1016/j.ajog.2020.04.031. Epub 2020 Apr 29. PMID 32360110
- [Background] Kovacevich GJ, Gaich SA, Lavin JP, Hopkins MP, Crane SS, Stewart J, Nelson D, Lavin LM. The prevalence of thromboembolic events among women with extended bed rest prescribed as part of the treatment for premature labor or preterm premature rupture of membranes. Am J Obstet Gynecol. 2000 May;182(5):1089-92. doi: 10.1067/mob.2000.105405. PMID 10819836